CLINICAL TRIAL: NCT05100186
Title: A Randomized, Controlled Study to Evaluate the Safety and Effectiveness of Treatment With an Intracanalicular Dexamethasone (0.4mg) Ophthalmic Insert in the Operating Room Following Cataract Surgery/Intraocular Lens Implant (IOL) Compared to Insertion 1-day Post-op - The SITE Study
Brief Title: The SITE Study - Dexamethasone Ophthalmic Insert In OR on Day of Surgery Versus In-office Post-Op Day 1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Joseph Kavanagh, MD (Other)
Responsible Party: Sponsor-Investigator, Joseph Kavanagh, MD, Principal Investigator, Eye Associates of South Texas
Organization: Eye Associates of South Texas (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SITE-2021-4002
Record Dates: First submitted 2021-10-15; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexamethasone Ophthalmic Insert (Experimental): Day of surgery, in OR placement versus Day 1 Post-Op, In-office (HOPD)
  Interventions: Drug: Dexamethasone 0.4 MG [Dextenza]

INTERVENTIONS:
Drug: Dexamethasone 0.4 MG [Dextenza] — Dextenza

SUMMARY:
To assess the safety and effectiveness of treatment with an intracanalicular dexamethasone (0.4mg) insert in the operating room following cataract surgery/intraocular lens implant (IOL) compared to insertion 1-day post-op.

DETAILED DESCRIPTION:
This is a randomized, controlled study to evaluate the safety and effectiveness of treatment with an intracanalicular dexamethasone (0.4mg) insert in the operating room following cataract surgery/intraocular lens implant (IOL) compared to insertion 1-day post-op.

There will be approximately 50 eyes with two groups:

Group 1 (up to 10 eyes) will receive the insert in the lower punctum on the day of surgery in the OR.

Group 2 (up to 40 eyes) will receive the insert in the lower punctum on the day after surgery in the HOPD.

Each subject's participation is expected to last for approximately 1 month and will be required to complete five scheduled visits over the course of the study period: Baseline (Screening Visit), Operative Visit/Insertion Day (Day 0), Day 1, Day 7 and Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for study participation if they:

  1. Are an adult subject aged 65 years or older
  2. Are planning to undergo non-complicated CCI CE/PCIOL in one or both eyes
  3. Are willing and able to comply with clinic visits and study related procedures
  4. Are willing and able to sign the informed consent form

Exclusion Criteria:

* Subjects are not eligible for study participation if they:

  1. Have active infectious systemic disease
  2. Have active infectious ocular or extraocular disease
  3. Have unobstructed nasolacrimal duct in the study eye(s)
  4. Have known hypersensitivity to dexamethasone or are a known steroid responder
  5. Have a history of ocular inflammation or macular edema
  6. Are currently being treated with immunomodulating agents in the study eye(s)
  7. Are currently being treated with immunosuppressants and/or oral steroids
  8. Are currently being treated with corticosteroid implant (i.e. Ozurdex)
  9. Have a history of herpes simplex virus keratitis or present active bacterial, viral, or fungal keratitis in either eye
  10. Have a history of complete punctal occlusion in one or both punctum
  11. Currently use topical ophthalmic steroid medications
  12. Are unwilling or unable to comply with the study protocol
  13. Are determined by the Investigator to not be included for reasons not already specified (e.g., systemic, behavioral, or other ocular disease/abnormality) or if the health of the subject or the validity of the study outcomes may be compromised by the subject's enrollment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Anterior Chamber Cells | Assessed on Day 7
  As measured by summed ocular inflammation score (0-4)
Ocular Pain | Assessed on Day 7
  As measured by ocular pain assessment numerical grading scale (0-10)

SECONDARY OUTCOMES:
Mean change in BCVA | Assessed on Day -1, Day 7, Day 30
  As measured by snellen VA
Percentage with complete absence of pain | Assessed on Day -1, Day 1, Day 7, Day 30
  As measured by ocular pain assessment numerical grading scale (0-10)
Percentage with complete absence of cell | Assessed on Day -1, Day 1, Day 7, Day 30
  As measured by summed ocular inflammation score (0-4)
Physician ease of insertion and visualization | Assessed on Day 1
  As measured by physician questionnaire